CLINICAL TRIAL: NCT01702870
Title: Comparison of Magnetic Resonance (MR) Imaging Against Clinical Criteria in the Diagnosis and Monitoring of Adult Idiopathic Myopathy
Brief Title: Diagnostic Accuracy of MR in Myositis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Warwick (Other)
Collaborators: West Midlands Comprehensive Local Research Network (Unknown); University Hospitals Coventry and Warwickshire NHS Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); The Royal College of Radiologists (Unknown)
Responsible Party: Principal Investigator, Dr. Terence Jones, Clinical Research Fellow in Radiology, University of Warwick
Other Study IDs: UoW-Myositis01
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Myositis; Muscular Disorders, Atrophic
Keywords: Magnetic resonance imaging
MeSH Terms: conditions — Myositis; Muscular Disorders, Atrophic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suspected myositis: Participants with suspected myositis based on clinical criteria (Bohan and Peters criteria) referred for Magnetic resonance imaging
  Interventions: Procedure: Magnetic Resonance Imaging
- Controls: Normal volunteers without myositis, who will undergo MR imaging to establish normal ranges of MR signal in health muscle
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging
  Other Names: Magnetic Resonance Imaging of the thighs

SUMMARY:
A prospective observational study to determine the effectiveness of magnetic resonance (MR) imaging in the diagnosis and monitoring of idiopathic myopathy in adult humans.

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies are a heterogeneous group of conditions characterised by skeletal muscle inflammation leading to proximal muscle weakness, often with tenderness, and occasionally dermatological manifestations. Diagnosis is clinical and is based on the Bohan and Peter criteria which comprises clinical examination, serological markers, electromyography (EMG) and muscle biopsy. This has relatively poor sensitivity and specificity. Muscle biopsy in particular has a false negative rate of 10-15% and is invasive. Clinical criteria also lack the discriminatory power to differentiate between recurrent (or breakthrough) myopathy and myopathy secondary to treatment with corticosteroid.

Magnetic resonance (MR) imaging has the advantage of being non-invasive, and is able to discriminate between different tissues, and to identify areas of inflammation. The aim of this study is to assess the effectiveness of MR sequences in the diagnosis of myopathy, monitoring of treatment response, and in differentiating between breakthrough myopathy and steroid-induced myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient referred for an MR scan with a suspected clinical diagnosis of myopathy.

Exclusion Criteria:

* Patient unable or unwilling to have an MR scan.
* Standard MR exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will be patients attendeing rheumatology outpoatient clinics with a suspected diagnosis of myopathy based on clinical criteria
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-11; Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
MR signal (T1w, T2w and STIR sequences) in muscle. | 2 years
  The correlation between MR signal and the clinical criteria will be measured

SECONDARY OUTCOMES:
Correlation between MR appearances (T1w, T2w and STIR signal on MR)and the symptom severity (Bohan and Peter criteria) | 2 years
Difference in MR signal between myopathy and steroid-induced myopathy, with sensitivity and specificity | 2 years

OTHER OUTCOMES:
Sensitivity and specificity of MR against the gold standard of clinical criteria | 2 years
  The MR signal will be compared against the Bohan and Peters criteria (the current gold standard) to determine sensitivity and specificity of the technique

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hutchinson, MD FRCR, Study Chair — Professor of Imaging (Radiology), University of Warwick; Terence Jones, MBChB FRCR, Principal Investigator — Clinical Research fellow in Radiology, University of Warwick
Locations (3):
- United Kingdom (3):
  - Salford Royal NHS Foundation Trust, Salford, Lancashire
  - George Eliot Hospital NHS Trust, Nuneaton, Warwickshire
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry, West Midlands